CLINICAL TRIAL: NCT03905629
Title: Validation of the Hospital Frailty Risk Score in Combination With Charlson/Elixhauser Comorbidity Coding Algorithms on French Hospital Databases
Brief Title: Validation of the Hospital Frailty Score in France
Acronym: HFRS France
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0018
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Elderly; Emergency Hospitalization; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 75 years and older hospitalized as an emergency: Patients considered will be all patients aged 75 years and older (on the day of the index admission) hospitalized as an emergency (i.e. after visit to ED) between january 2017 and december 2017.
  Interventions: Other: None (retrospective observational study)

INTERVENTIONS:
Other: None (retrospective observational study) — This multi-centric retrospective observational cohort study is conducted using the PMSI. Predictive ability of HFRS estimated on the basis of 3 binary outcomes: 30-day in-patient mortality (main outcome), 30-day emergency and potentially avoidable readmission, length of stay >15 days. Odds ratios (ORs) and c-statistics calculated and compared to the original UK results in order to validate the use of the HFRS in France. Other secondary objectives include:
  * Evaluate agreement between HFRS and Charlson or Elixhauser comorbidity indices
  * Evaluate ability of HFRS combined with comorbidity indices (Charlson on one hand, and Elixhauser on other hand), to predict 30-day in-patient mortality, 30-day emergency and potentially avoidable readmissions, and long length of stay
  * Identify specific risk associations in France of a high risk of frailty (as assessed by the HFRS) with individual, organizational and territorial factors
  Other Names: Validation of the HFRS in Combination With Charlson/Elixhauser Comorbidity Coding Algorithms on the French national PMSI database

SUMMARY:
Older people are increasing users of health care globally. Constraints in bed capacity and resources raise important challenges with regards to management of older people with complex needs, which usually require assertive and holistic assessment. It is important, therefore, to identify aged patients most likely to benefit from such frailty-attuned approaches of care. A previous study using national Hospital Episodes Statistics conducted in the United Kingdom (UK) showed that patients aged over 75 years with characteristics of frailty and at risk of adverse health-care outcomes can be identified using routinely collected data (Gilbert T et al., Lancet 2018). This study lead to the development of the Hospital Frailty Risk Score (HFRS), which is based on International Statistical Classification of Diseases and Related Health Problems 10 (ICD-10) diagnosis codes and has the potential to be used in other countries worldwide, using the ICD-10 coding framework, to identify patients at risk of frailty at the hospital and commissioners levels, as well as for database research purposes. This score has successfully been validated in Canada, Australia and Switzerland. The aim of the present study is to evaluate the ability of the HFRS to predict 30-day in-patient mortality of patients aged 75 years and older admitted to French hospitals as an emergency.

ELIGIBILITY:
Inclusion Criteria:

* age 75 years or over (on the day of the index admission)
* hospitalized as an emergency (i.e. after visit to ED)

Exclusion Criteria:

* none

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients considered will be all patients aged 75 years and older hospitalized as an emergency over a one year period ranging from January to December 2017.
  According to a preliminary extraction, we expect to include approximately one million patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
30-day in-patient mortality | In-patient mortality within 30 days from admission (index hospitalization)
  The main outcome measure will be 30-day in-patient mortality. Mortality data will be limited to in-hospital mortality, which will be directly available from the PMSI database.

CONTACTS AND LOCATIONS:
Locations (1):
- service de court séjour gériatrique, Hôpital Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Derived] Gilbert T, Cordier Q, Polazzi S, Bonnefoy M, Keeble E, Street A, Conroy S, Duclos A. External validation of the Hospital Frailty Risk Score in France. Age Ageing. 2022 Jan 6;51(1):afab126. doi: 10.1093/ageing/afab126. PMID 34185827